CLINICAL TRIAL: NCT01410019
Title: Protocol No. 2 of Gene Therapy for X-linked Severe Combined Immunodeficiency (SCID-X1) Using a Self Retroviral Vector - SCID2
Brief Title: Gene Therapy for X-linked Severe Combined Immunodeficiency
Acronym: SCID2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P071204; 2008-002380-14 (EudraCT Number)
Record Dates: First submitted 2011-06-21; First posted 2011-08-04 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: X-linked Severe Combined Immunodeficiency
Keywords: X-linked Severe Combined Immunodeficiency (SCID-X1); severe infection; gene therapy; HLA identical family donor; without HLA identical unrelated donor
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases; Infections | interventions — Genetic Engineering

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Gene transfer
  Interventions: Other: Gene transfer

INTERVENTIONS:
Other: Gene transfer — Single infusion of autologous CD34+ cells transduced with the self-inactivating (SIN) GAMMARETROVIRAL vector pSRS11.EFS.IL2RG.pre

SUMMARY:
X-linked severe combined immunodeficiency (SCID-X1) is an inherited disorder that results in failure of development of the immune system in boys. This trial aims to treat SCID-X1 patients using gene therapy to replace the defective gene.

DETAILED DESCRIPTION:
The objective of this protocol is to reinitiate an ex vivo gene therapy clinical protocol to treat patients with SCID-X1 without HLA identical family donor nor HLA identical unrelated donor (bone marrow and cord blood) available in an adequate time with the clinical conditions of the patient at diagnosis (approximately 6 weeks). This clinical protocol No. 2 of SCID-X1 must be as efficient than the previous one but must involve a risk of insertional mutagenesis significantly reduced as compared to the first protocol.

The main purpose of the study is the study of toxicity: tolerance and incidence of serious adverse effects.

Secondary goals are the evaluation of immune reconstitution allowing the cure of infections present at the time of gene therapy, assessment of integration sites, and finally the long-term correction of immunosuppression.

1. safety assessment : clinical effects, possible emergence of clonal lymphocyte proliferation, potential activation of proto-oncogene;
2. efficacy assessment of ex vivo transduction of CD34 + hematopoietic stem cells of the patient through the use of retroviral vector pSRS11.EFS.IL2RG.pre;
3. assessment of immune reconstitution : phenotype, number and function of different T, NK and B cells subpopulations;
4. longitudinal evaluation of clinical effects in terms of improvement or complete restoration of immunity;
5. biological efficacy assessment of this new vector SIN, assessment of molecular characteristics of retroviral integration.

ELIGIBILITY:
Inclusion criteria :

* Boys diagnosed during the first year of life
* Diagnosis of classical SCID-X1 based on immunophenotype (absent, or reduced numbers of non-functional T lymphocytes) and confirmed by DNA sequencing
* No HLA identical family donor and no HLA identical unrelated donor (10/10 antigens) found in the 6 weeks following the beginning of the search. This period could be shortened if the probability to find a donor is low or if the clinical situation (gravity) required
* Presence of a severe infection: pneumonitis and / or chronic diarrhea, or infection with herpes viruses or parainfluenza type 3 or adenovirus, or disseminated BCG infection, or presence of severe diarrhea and a severe compromise of the general state with denutrition
* Or failure of a HLA HAPLO-identical bone marrow transplant within 10 years after transplantation
* In all cases:

  * No family background of cancer in childhood.
  * No cytogenetic abnormalities (medullary karyotype) and no detection of main rearrangements associated with acute leukemia of children
  * Parental/guardian voluntary consent

Exclusion criteria :

* Atypical health with autologous T> 500/ml3
* Infection by HIV 1 or 2
* Allogeneic HSC completed (excluding situations of failure)
* Existence of an HLA identical family donor or HLA identical unrelated donor
* No severe infections in a child with a preserved general state
* Family background of cancer in childhood
* Detection of cytogenetic abnormality and / or rearrangement associated with acute leukemia of children
* No affiliation to a social security scheme (beneficiary or assignee)

Max Age: 12 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2010-12; Primary Completion 2015-06-16 (Actual); Study Completion 2015-06-16 (Actual)

PRIMARY OUTCOMES:
Assessment of immunological reconstitution at short term | month 4
  T cells proliferation T cells and B cells repertory by immunofluorescence T, NK and B Lymphocytes phenotyping Immunoglobulins dosage IgG, A, M, E and antibody production

SECONDARY OUTCOMES:
Molecular characterization of gene transfer | every 15 days during 3 months, once per month until 6 months, every 3 months until year 1, every year until year 10
  PCR of vector
Analysis of activated proto-oncogene s expression | every 4 months during 2 years and every 6 months indefinitely
  Immunofluorescence analysis of the relative expression of different families of TCR alpha beta et gamma delta LAM PCR analysis and sequencing of integration sites

CONTACTS AND LOCATIONS:
Overall Officials: Alain Fischer, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Necker, Paris, France

REFERENCES:
- [Background] Hacein-Bey-Abina S, Pai SY, Gaspar HB, Armant M, Berry CC, Blanche S, Bleesing J, Blondeau J, de Boer H, Buckland KF, Caccavelli L, Cros G, De Oliveira S, Fernandez KS, Guo D, Harris CE, Hopkins G, Lehmann LE, Lim A, London WB, van der Loo JC, Malani N, Male F, Malik P, Marinovic MA, McNicol AM, Moshous D, Neven B, Oleastro M, Picard C, Ritz J, Rivat C, Schambach A, Shaw KL, Sherman EA, Silberstein LE, Six E, Touzot F, Tsytsykova A, Xu-Bayford J, Baum C, Bushman FD, Fischer A, Kohn DB, Filipovich AH, Notarangelo LD, Cavazzana M, Williams DA, Thrasher AJ. A modified gamma-retrovirus vector for X-linked severe combined immunodeficiency. N Engl J Med. 2014 Oct 9;371(15):1407-17. doi: 10.1056/NEJMoa1404588. PMID 25295500
- [Background] Cavazzana-Calvo M, Hacein-Bey S, de Saint Basile G, Gross F, Yvon E, Nusbaum P, Selz F, Hue C, Certain S, Casanova JL, Bousso P, Deist FL, Fischer A. Gene therapy of human severe combined immunodeficiency (SCID)-X1 disease. Science. 2000 Apr 28;288(5466):669-72. doi: 10.1126/science.288.5466.669. PMID 10784449
- [Background] Hacein-Bey-Abina S, Le Deist F, Carlier F, Bouneaud C, Hue C, De Villartay JP, Thrasher AJ, Wulffraat N, Sorensen R, Dupuis-Girod S, Fischer A, Davies EG, Kuis W, Leiva L, Cavazzana-Calvo M. Sustained correction of X-linked severe combined immunodeficiency by ex vivo gene therapy. N Engl J Med. 2002 Apr 18;346(16):1185-93. doi: 10.1056/NEJMoa012616. PMID 11961146
- [Background] Hacein-Bey-Abina S, Hauer J, Lim A, Picard C, Wang GP, Berry CC, Martinache C, Rieux-Laucat F, Latour S, Belohradsky BH, Leiva L, Sorensen R, Debre M, Casanova JL, Blanche S, Durandy A, Bushman FD, Fischer A, Cavazzana-Calvo M. Efficacy of gene therapy for X-linked severe combined immunodeficiency. N Engl J Med. 2010 Jul 22;363(4):355-64. doi: 10.1056/NEJMoa1000164. PMID 20660403
- [Derived] Clarke EL, Connell AJ, Six E, Kadry NA, Abbas AA, Hwang Y, Everett JK, Hofstaedter CE, Marsh R, Armant M, Kelsen J, Notarangelo LD, Collman RG, Hacein-Bey-Abina S, Kohn DB, Cavazzana M, Fischer A, Williams DA, Pai SY, Bushman FD. T cell dynamics and response of the microbiota after gene therapy to treat X-linked severe combined immunodeficiency. Genome Med. 2018 Sep 28;10(1):70. doi: 10.1186/s13073-018-0580-z. PMID 30261899